CLINICAL TRIAL: NCT02909309
Title: Pilot Study : Evaluation of a Mandibular and Abdominal Motion Detection Sensors (JAWAC) to Prevent Apnea During Sedation With Propofol in TCI Mode
Brief Title: Pilot Study : New Sensors to Monitor Apnea During Sedation
Acronym: JAWAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Luc Barvais, Professor and head of the cardiothoracic and vascular anesthesia Clinics, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P2016/329
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Sleep Apnea, Obstructive; Anesthesia
Keywords: Propofol; Deep Sedation; Anoxia; Hypercapnia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypoxia; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALL INCLUDED PATIENTS (Other): A single arm for this study. All the patients benefit of both systems. The participants are their own control.
  Non invasive sensors are used to monitor and record data of those two systems in a synchron way ( JAWAC / Capnoline + Spo2).
  Interventions: Device: JAWAC system + Capnoline + Spo2

INTERVENTIONS:
Device: JAWAC system + Capnoline + Spo2 — measure mandibular mouvements + etCO2 + pulse oxymetry, respectively

SUMMARY:
Evaluation of a Mandibular and Abdominal Motion Detection Sensor (JAWAC) to Prevent Apnea During Sedation With Propofol in TCI Mode

DETAILED DESCRIPTION:
In 2016 , monitoring of propofol sedation , currently recommended by the American Society of Anaesthesiology and European companies includes among others, a pulse oximeter (SpO2) and a continuous measurement of CO2 exhaled by an appropriate device (CapnoLine). This monitoring does not allow to anticipate the occurrence of obstructive apnea .

The anticipation of the occurrence of apnea or airway obstruction using this type of monitoring could allow the anesthesiologist to act earlier on the titration of propofol and maintaining the airway. This would avoid the side effects associated with hypoxemia and hypercapnia and therefore further improve patient safety .

This pilot study tests the JAWAC system to detect those apneas.

This is an interventional diagnostic study on the JAWAC monitoring system validation in a prospective cohort of patients undergoing sedation in order to provoke sleep apnea. Indeed , sedation technique is already used with propofol during snoring provocation tests in patients at risk for sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient scheduled for a sleep apnea provocation test under sedation by propofol
* Hospital Erasme during the period of the study.

Exclusion Criteria:

1. Patient Refusal
2. Patient Age: 18 years and under 80 years
3. Intervention earlier in the mandible or thorax
4. A history of facial burn
5. Allergy tape

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Optimal JAWAC signal threshold detecting obstructive apnea | at time of anesthesia
  The apnea is defined clinically by the anesthesiologist with the help of the capnoLine/Spo2. The purpose is to define the optimal signal detection during a continuous record of the system JAWAC associated with the occurrence of obstructive apnea.
  The results will give a variation in centimeters for a certain amount of time. It is possible that the optimal signal detection will be a combination of different sensors.
  The sensibility, specificity versus precocity of the signal will be studied.

SECONDARY OUTCOMES:
Time limit between the detection of each system and the episode of désaturation | at time of anesthesia
  The assumption is that the signal JAWAC enable an earlier response of the anesthetist and a priori reduce the occurrence of desaturation at the onset of obstructive apnea compared to the capnoLine/spo2 system.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Barvais, Study Director — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tinker JH, Dull DL, Caplan RA, Ward RJ, Cheney FW. Role of monitoring devices in prevention of anesthetic mishaps: a closed claims analysis. Anesthesiology. 1989 Oct;71(4):541-6. doi: 10.1097/00000542-198910000-00010. PMID 2508510
- [Background] Senny F, Destine J, Poirrier R. Midsagittal jaw movement analysis for the scoring of sleep apneas and hypopneas. IEEE Trans Biomed Eng. 2008 Jan;55(1):87-95. doi: 10.1109/TBME.2007.899351. PMID 18232350
- [Background] Niklewski PJ, Phero JC, Martin JF, Lisco SJ. A novel index of hypoxemia for assessment of risk during procedural sedation. Anesth Analg. 2014 Oct;119(4):848-856. doi: 10.1213/ANE.0000000000000371. PMID 25232693
- [Derived] Ponthieu N, Coeckelenbergh S, Engelman E, Tuna T, Van Obbergh L, Barvais L. Synchronized mandibular movement and capnography: a novel approach to obstructive airway detection during procedural sedation-a post hoc analysis of a prospective study. J Clin Monit Comput. 2019 Dec;33(6):1065-1070. doi: 10.1007/s10877-018-00250-3. Epub 2019 Jan 4. PMID 30610518